CLINICAL TRIAL: NCT04321512
Title: Study of Circulating Monocytes in Patients With Ischemic Vascular Disease
Status: Recruiting | Type: Observational
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Bruce Liang, Professor of Medicine, Director Pat and Jim Calhoun Cardiovascular Center, UConn Health
Other Study IDs: 13-119-2
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Myocardial Infarction; Stroke, Ischemic; Ischemia
MeSH Terms: conditions — Myocardial Infarction; Ischemic Stroke; Ischemia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum, whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: There is no intervention given to the subjects — Not appicable

SUMMARY:
The purpose of this research study is to discover the functions of circulating white blood cells, called monocytes, and associated circulating substances in heart attack and ischemic stroke patients. Ischemic Strokes (clots) occur as a result of an obstruction within a blood vessel supplying blood to the brain. A type of monocyte carrying a surface marker called "P2X4" helps the immune system sense and respond to danger signals from the body such as heart muscle and brain tissue injuries.

The researchers expect to learn more about how these monocyte cells react to heart and brain tissue injury, and how the cells may then produce proteins or other chemical substances which promote the healing of heart muscle after heart attack and brain tissue after an ischemic stroke.

DETAILED DESCRIPTION:
The research objective here is to perform a pilot study in determining the level of such monocytes in MI/stroke patients at various times after the acute ischemic event. As controls, both stable coronary disease and healthy control subjects will be enrolled in whom these circulating cells will be determined.

The research objective will be accomplished via the following specific aim:

The specific aim will determine the levels of P2X4 monocytes, Flt-1/VEGFR-1 and CD13 monocytes. The researchers may collect three blood samples at various time points. The samples will be collected within 48 hours of admission to the hospital, 2-14, and 30-120 days following MI/stroke. As a control, levels of P2X4, Flt-1+ (VEGFR-1+) and CD13 monocytes in age- matched healthy subjects and in SCAD subjects will be used. Additionally for CD13 monocytes, the researchers plan to test if CD13 is phosphorylated in the circulating monocytes of patients who have undergone myocardial/cerebral infarction and determine its utility as a biomarker of infarct size.

Although the study is not designed to determine whether those MI/stroke patients within the top quartile of P2X4 or Flt-1+ (VEGFR-1+) or CD13 monocyte levels are more prone to develop severe tissue or organ dysfunction, the study will collect baseline and subsequent clinical data set and should position the study team to test this hypothesis in the future.

The researchers might expect to show that MI/stroke patients have a higher level of P2X4, Flt-1+ (VEGFR-1+) and/or CD13 monocytes as well as circulating cytokines and metabolites as compared to SCAD and age-matched healthy controls. The researchers might also expect that thrombectomy samples from ischemic stroke patients will have higher inflammatory cytokines and inflammatory monocytes.

Objectives:

* To obtain blood samples from STEMI patients for determination of P2X4, Flt-1+ (VEGFR-1+) and CD13 monocyte levels as well as circulating cytokines and metabolites on the days: 1(within 48 hours of admission), 2-14, and 30-120 days after the MI.
* To obtain blood samples from NSTEMI (non-ST segment elevation MI) patients for determination of P2X4, Flt-1+ (VEGFR-1+) and CD13 monocyte levels as well as circulating cytokines and metabolites on the days: 1(within 48 hours of admission hospital), 2-14, and 30-120 days after the MI.
* To obtain blood samples from ischemic stroke patients for determination of P2X4, Flt-1+ (VEGFR-1+) and CD13 monocyte levels as well as circulating cytokines and metabolites on the days: 1(within 48 hours of admission), 2-14, and 30-120 days after the ischemic event. In addition, thrombectomy samples which are normally discarded, when obtained and available, will be used.
* To obtain blood samples from age-matched SCAD and healthy control subjects for a one-time determination of P2X4, Flt-1+ (VEGFR-1+) and CD13 monocyte as well as circulating cytokines and metabolites levels.
* To compare the levels in STEMI, NSTEMI and ischemic stroke vs. those of SCAD and healthy control subjects.

Hypotheses:

STEMI, NSTEMI and stroke subjects will have a higher level of P2X4, Flt-1+ (VEGFR- 1+) and CD13 monocytes than age-matched SCAD and healthy control subjects.

ELIGIBILITY:
Inclusion Criteria:

* STEMI Patients: Men and women aged 18 years and over, with symptoms, physical signs and ECG changes characteristic of STEMI.
* NSTEMI Patients: Men and women aged 18 years and over, with symptoms, physical signs and ECG changes characteristic of NSTEMI.
* Stable CAD Patients: men and women aged 18 years and older with coronary artery disease proven by prior MI history, angiography or stress test but without any unstable angina or acute coronary syndrome.
* Ischemic Stroke Patients: Men and women aged 18 years and over, with symptoms, physical signs and CT/MRI changes characteristic of ischemic stroke.
* Healthy Controls: Men and women aged 18 years and over, without heart failure, coronary disease, hypertension, diabetes or other chronic diseases. Control subjects will be recruited from within the community of UConn Health via advertisement.

Exclusion Criteria:

* Subjects who are unable to give informed consent (with the exception of the ischemic stroke arm patients, see Protocol Design below) and pregnant subjects.
* Subjects who had any history of embolic, ischemic or hemorrhagic stroke within the last 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment will take place at UConn Health Center. The target populations of 300 will be those with STEMI (60 subjects), NSTEMI (60 subjects) and SCAD (60 subjects), ischemic stroke (60 subjects), and age-matched non-disease subjects (60 subjects). The researchers anticipate that 5% of all recruited subjects will be African American and another 3% will be Latinos and Asians. This represents the distribution of populations recruited in the past for heart disease studies.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-12-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Hospitalization for Myocardial Infarction, Stroke, or death | 3 years
  myocardial infarction, stroke or death

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Liang, MD, Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No